CLINICAL TRIAL: NCT05215483
Title: Availability and Advice on Test Uptake During the COVID-19 Pandemic: a Vignette Study on Lateral Flow Testing Policy in the Netherlands.
Brief Title: Availability and Advice on Test Uptake During the COVID-19 Pandemic: a Vignette Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Principal Investigator, Colene Zomer, Researcher Corona Behavioural Unit, National Institute for Public Health and the Environment (RIVM)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: G&M-537
Record Dates: First submitted 2022-01-24; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: Test intentions; Lateral Flow test uptake
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: In an online randomised multi-factorial survey (vignette study) participants are randomised to assess four scenario's. Between subject testing advise is randomised (IV1; 2 levels) and the availability of LFT (IV2; 2 levels). Within subject we asked participants to assess their most likely behaviour on day 1 of symptoms and day 3 of unchanged symptoms (IV3; 2 levels). Corona-related symptoms are randomly presented (IV4; 4 levels) and new incidences of symptoms are presented in additional vignettes describing new months (IV5; 4 levels).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Customised advice + LFT available at home (Experimental): Respondents will see an altered testing advice in text and picture in which they are allowed to use LFT with corona related symptoms.
  Respondents will informed in writing that they don't currently have any LFT available at home.
  Interventions: Behavioral: Customised testing advice; Behavioral: LFT available
- Customised advice + No LFT available at home (Experimental): Respondents will see an altered testing advice in text and picture in which they are allowed to use LFT with corona related symptoms.
  Respondents will informed in writing that they don't currently have any LFT available at home.
  Interventions: Behavioral: Customised testing advice; Behavioral: No LFT available
- Regular advice + LFT available at home (Experimental): Respondents will see the regular testing advice in text and picture with the current governmental advice to visit a test facility with corona related symptoms.
  Respondents will informed in writing that they don't currently have any LFT available at home.
  Interventions: Behavioral: Regular testing advice; Behavioral: LFT available
- Regular advice + No LFT available at home (Active Comparator): Respondents will see the regular testing advice in text and picture with the current governmental advice to visit a test facility with corona related symptoms.
  Respondents will informed in writing that they don't currently have any LFT available at home.
  Interventions: Behavioral: Regular testing advice; Behavioral: No LFT available

INTERVENTIONS:
Behavioral: Customised testing advice — Customised advice: With Corona related symptoms, get tested at a test facility. If this isn't possible, use a Lateral Flow test.
  Arms: Customised advice + LFT available at home; Customised advice + No LFT available at home
Behavioral: Regular testing advice — Government guideline testing advice: "With Corona related symptoms, get tested at a test facility".
  Arms: Regular advice + LFT available at home; Regular advice + No LFT available at home
Behavioral: LFT available — LFT availability: Enough lateral flow tests available at home
  Arms: Customised advice + LFT available at home; Regular advice + LFT available at home
Behavioral: No LFT available — LFT availability: No lateral flow tests available at home
  Arms: Customised advice + No LFT available at home; Regular advice + No LFT available at home

SUMMARY:
Lateral Flow Testing (LFT) use for COVID-19 related symptoms continues to rise, despite governmental advice to test at a test facility. In this study we investigate whether 1) adjusting the governmental testing advice will lead to a collective increase of people who test with COVID-19 symptoms and if this leads to a higher strategy sensitivity.

DETAILED DESCRIPTION:
In an online randomised multi-factorial survey (vignette study) participants are randomised to assess four scenario's. Between subject testing advise is randomised (IV1; 2 levels) and the availability of LFT (IV2; 2 levels). Within subject we asked participants to assess their most likely behaviour on day 1 of symptoms and day 3 of unchanged symptoms (IV3; 2 levels). Corona-related symptoms are randomly presented (IV4; 4 levels) and new incidences of symptoms are presented in additional vignettes describing new months (IV5; 4 levels).

Subjects are asked to immerse themselves in the scenario's before answering what their most likely behaviour would be: a) go to a test facility b) use a LFT c) wait and see or 4) no test. Participants who didn't choose the test facility on day 1 were presented with the same vignette on day 3 with unchanged symptoms, and were asked their most likely behaviour again.

After assessing the scenario's, participants fill in a questionnaire assessing demographics, behavioural determinants related to test behaviour, vaccine status, current symptoms and previous experience with Corona and testing.

The primary outcomes is defined as the average strategy sensitivity over time and therefore the chance of detecting a Covid-infection. Average strategy sensitivity is calculated by converting the choice of testing behaviour into the corresponding sensitivity score (PCR =1, LFT day 1 = .8, LFT day 3 = .7, wait and see and no test = 0), averaged over four scenario's.

Our primary hypothesis is:

1. Adjusting the governmental testing advice will lead to a higher strategy sensitivity.

   In follow-up analysis we will explore the following hypothesis:
2. Availability of LFT at home will lead to a higher strategy sensitivity.
3. The type of corona related symptoms (mild or severe) are predictive of the type of test used.
4. When confronted with a new incidence of corona-related symptoms over time, strategy sensitivity will decline.

ELIGIBILITY:
Participants were recruited from an online research panel representative for the Dutch population.

Inclusion Criteria:

* non

Exclusion Criteria:

* non

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3270 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Average strategy sensitivity over time: day 1 | average strategy sensitivity day 1
  The sensitivity of the test chosen was used to convert each answer: test facility on day 1 = 1, LFT on day 1= 0.8, Wait and see or No test = 0. Sensitivity scores were then averaged over the four scenario's.
Maximum average strategy sensitivity over time | maximum average strategy sensitivity day 1 and 3
  The sensitivity of the test chosen was used to convert each answer: test facility on day 1 or day 3 = 1, LFT on day 1= 0.8, LFT on day 3= 0.7, Wait and see or No test = 0. Sensitivity scores were then averaged over the four scenario's. The highest score of day 1 and day 3 was used to calculate the maximum sensitivity score.

SECONDARY OUTCOMES:
Willingness to test day 1 | Day 1
  Willingness to test on day 1 (LFT & PCR =1, no test = 0), averaged over the four scenario's.
Willingness to test - maximum | Day 1 and 3
  Willingness to test on day 1 and 3 (LFT & PCR =1, no test = 0), averaged over the four scenario's.
Type of test chosen day 1 | Day 1
  Percentage of testing behaviour (test facility, LFT, Wait and see, No test) on day 1, averaged over the four scenario's.
Type of test chosen day 3 | Day 3
  Percentage of testing behaviour (test facility, LFT, Wait and see, No test) on day 3, averaged over the four scenario's.

CONTACTS AND LOCATIONS:
Overall Officials: Marijn de Bruin, prof, Study Chair — RIVM
Locations (1):
- National Institute for Public Health and the Environment, Bilthoven, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Do members of the public think they should use lateral flow tests or PCR tests when they have COVID-19-like symptoms? The COVID-19 Rapid Survey of Adherence to Interventions and Responses [CORSAIR] study, — https://doi.org/10.1016/j.puhe.2021.07.023